CLINICAL TRIAL: NCT00467558
Title: A Double-Blind, Placebo-Controlled Study of Naltrexone in Compulsive Sexual Behavior
Brief Title: Double-Blind Naltrexone in Compulsive Sexual Behavior
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0701M00804
Record Dates: First submitted 2007-04-27; First posted 2007-04-30 (Estimated); Results first posted 2012-05-18 (Estimated); Last update posted 2012-05-18 (Estimated); Status verified 2012-04

CONDITIONS: Compulsive Sexual Behavior
Keywords: Impulse Control Disorder; Compulsive Sexual Behavior
MeSH Terms: conditions — Compulsive Sexual Behavior Disorder; Disruptive, Impulse Control, and Conduct Disorders | interventions — Naltrexone; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Naltrexone (Active Comparator): Naltrexone 50mg-150mg by mouth per day.
  Interventions: Drug: Naltrexone
- Placebo (Placebo Comparator): Placebo pills (1-3 pills daily) depending upon dose prescribed by study physician
  Interventions: Drug: Sugar pill

INTERVENTIONS:
Drug: Naltrexone — daily
  Other Names: Revia
  Arms: Naltrexone
Drug: Sugar pill — daily
  Arms: Placebo

SUMMARY:
The goal of the proposed study is to evaluate the efficacy and safety of naltrexone in compulsive sexual behavior. Twenty subjects with DSM-IV compulsive sexual behavior will receive 8 weeks of naltrexone or placebo. The hypothesis to be tested is that naltrexone will be effective in reducing the urges to act out sexually in patients with compulsive sexual behavior. The proposed study will provide needed data on the treatment of a disabling disorder that currently lacks a clearly effective treatment.

DETAILED DESCRIPTION:
The proposed study will consist of 8 weeks of treatment with either naltrexone or placebo in 20 subjects with compulsive sexual behavior.

ELIGIBILITY:
Inclusion Criteria:

1. men and women age 21-75;
2. current diagnosis of compulsive sexual behavior

Exclusion Criteria:

1. unstable medical illness or clinically significant abnormalities on prestudy laboratory tests or physical examination;
2. history of seizures;
3. myocardial infarction within 6 months;
4. current pregnancy or lactation, or inadequate contraception in women of childbearing potential;
5. clinically significant suicidality;
6. current or recent (past 1 month) DSM-IV substance abuse or dependence;
7. illegal substance within 2 weeks of study initiation;
8. initiation of psychotherapy or behavior therapy from a mental health professional within 3 months prior to study baseline;
9. initiation of a psychotropic medication within 2 months prior to study inclusion;
10. previous treatment with naltrexone; and
11. treatment with investigational medication or depot neuroleptics within 3 months, with fluoxetine within 6 weeks, or with other psychotropics within 2 weeks prior to study baseline

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon E Grant, M.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Naltrexone | Placebo
Started | 4 | 3
Completed | 2 | 3
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naltrexone | Placebo | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 7
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 27.67 (7.37) | 35.67 (10.69) | 31.87 (9.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 7

OUTCOME MEASURES:

1. Secondary Outcome: Clinical Global Impression Scale - Severity
Description: The CGI consists of two reliable and valid 7-item Likert scales used to assess severity in clinical symptoms. The scale ranges from 1 = "very much improved" to 7 = "very much worse." The CGI severity scale was used at each visit and ranges from 1 = "not ill at all" to 7 = "among the most extremely ill."
Time Frame: Assessed at each visit (every two weeks) until participation in the study was done (Week 8)
Population: Reported scores are Mean and standard deviation for Subjects last visit (Week 8 or last-observation carried forward).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 3 | 3
units on a scale | 2.33 (1.53) | 2.67 (0.58)

2. Primary Outcome: Yale Brown Obsessive Compulsive Scale Modified for Compulsive Sexual Behavior (YBOCS)
Description: The YBOCS is a reliable and valid, 10-item, clinician-administered scale that rates buying symptoms within the last seven days, on a severity scale from 0 to 4 for each item (total scores range from 0 to 40 with higher scores reflecting greater illness severity).
Time Frame: Assessed at each visit (every two weeks) until participation in the study was done (Week 8)
Population: Reported scores are Mean and standard deviation for Subjects last visit (Week 8 or last-observation carried forward).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Naltrexone | Placebo
Number analyzed (Participants) | 3 | 3
units on a scale | 8 (7) | 9.33 (1.15)

ADVERSE EVENTS:
Arm/Group | Naltrexone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 0/4 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No